CLINICAL TRIAL: NCT06367686
Title: Detecting Systemic Carbon Dioxide Levels With a Novel Biosensor; The DISCO-study
Brief Title: Detecting Systemic Carbon Dioxide Levels With a Novel Biosensor
Acronym: DISCO
Status: Recruiting | Type: Observational
Sponsor: The Hospital of Vestfold (Other)
Collaborators: Sensocure AS (Industry)
Responsible Party: Principal Investigator, Anne-Marie Gabrielsen, Senior consultant, The Hospital of Vestfold
Other Study IDs: REK KULMU B 714179
Record Dates: First submitted 2024-03-05; First posted 2024-04-16 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hypercapnic Respiratory Failure; Pulmonary Disease, Chronic Obstructive; Neuromuscular Diseases; Obesity Hypoventilation Syndrome (OHS)
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Neuromuscular Diseases; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chronic obstructive pulmonary disease: 3 Chronic obstructive pulmonary disease patients monitored with IscAlert sensor at nasal mucosa for 8-14 hours during the night
  Interventions: Device: IscAlert sensor
- Neuromuscular disease: 3 Neuromuscular disease patients monitored with IscAlert sensor at nasal mucosa for 8-14 hours during the night
  Interventions: Device: IscAlert sensor
- Obesity hypoventilation syndrome: 3 Obesity hypoventilation syndrome patients monitored with IscAlert sensor at nasal mucosa for 8-14 hours during the night
  Interventions: Device: IscAlert sensor
- Healthy volunteers: 2 healthy volunteers monitored with IscAlert sensor at nasal mucosa for approximately 8 hours during daytime
  Interventions: Device: IscAlert sensor

INTERVENTIONS:
Device: IscAlert sensor — Insertion of an IscAlert sensor at the nasal mucosa

SUMMARY:
The study is an open, prospective, single center clinical observational pilot investigation. The aim is to compare the carbon dioxide values measured by the IscAlert sensor, which is inserted in proximity to the nasal mucosa. The study wants to investigate if the nasal mucosa application and measurements are feasible, what kind of possible complications such a measurement can cause, and if the measurements can be a surrogate marker for systemic carbon dioxide values.

DETAILED DESCRIPTION:
he study is an open, prospective, single center clinical observational pilot investigation including 9 patients and 2 healthy volunteers. The aim is to compare the carbon dioxide values measured by the IscAlert sensor, which is inserted in proximity to the nasal mucosa, with the transcutaneous carbon dioxide values measured at the forehead by a transcutaneous carbon dioxide-monitor, the arterial carbon dioxide measurements performed by blood gas analyses, and carbon dioxide measurements registered with the IscAlert sensor implanted in the muscle of the forearm. The study wants to investigate if the nasal mucosa application and measurements are feasible, what kind of possible complications such a measurement can cause, and if the measurements can be a surrogate marker for systemic carbon dioxide values. The study will include patients with a tendency to hypoventilation, thereby giving rise to a carbon dioxide retention; 3 patients with chronic obstructive pulmonary disease with suspected hypercapnic respiratory failure who are evaluated for non-invasive mask-treatment and long-term oxygen treatment supply if needed. 3 patients with neuromuscular disorders and 3 patients with obesity hypoventilation syndrome who are evaluated for non-invasive mask treatment. The measurements will last for about 8 to 14 hours at night while the patients are sleeping. In addition, the study will also include 2 healthy volunteers as a control group. They will have the equipment mounted on them for about 8 hours during the day in connection with normal office work. Follow up by telephone 7 days +/-2 days after the measurements are finished. The inclusion period is expected to be about 9 months.

ELIGIBILITY:
Inclusion Criteria:

The subject must meet all of the following inclusion criteria at the time of enrolment:

EITHER

1. Patient are at risk of hypoventilation and thus carbon dioxide retention.
2. Either

   1. Under evaluation for treatment with non-invasive ventilation and maybe Long term oxygen treatment due to chronic obstructive pulmonary disease or
   2. Under evaluation for non-invasive ventilation support due to Obesity hypoventilation syndrome or due to a neuromuscular disorder.

   OR
3. Healthy volunteers

   ALL subjects:
4. Subject must be 18 years or older
5. Subject must be able to give written informed consent

Exclusion Criteria:

1. Known allergy to local anesthetics.
2. Participants should not have any kind of (direct or indirect) affiliation to Sensocure AS
3. Healthy volunteers: No heart-, lung-, or circulatory diseases, no bleeding disorder, no sleep disorders
4. Healthy volunteers should not have any kind of (direct or indirect) acquaintanceship to the investigators
5. Active smoker/use of snuff

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Nine patients will be selected consequtive from the hypoventilation assessment planning program at the site. Additionally, two healthy individuals, who have no heart-, lung-, or circulatory diseases, no bleeding disorder, no sleep disorders, and no ties whatsoever to the sponsor (Sensocure AS), will be included as volunteers. Otherwise completely freely chosen by the investigators except they must not have any kind of (direct or indirect) acquaintanceship to the investigators. Eligible subjects will be invited to participate in this clinical investigation. All the subjects will be included at least one day before study procedure starts.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Partial pressure (level) of carbon dioxide at the nasal mucosa | 14 hours
  Nasal mucosa's partial pressure of carbon dioxide (kPa) during insertion period

SECONDARY OUTCOMES:
Bleeding | 7 days
  Amount of blood from insertion site (ml)
Infection | 7 days
  Infection from insertion site at the discretion of the investigator (yes or no)
Sinusitis | 7 days
  Developement of sinusitis at the discretion of the investigator (yes or no)
Ulceration | 7 days
  Developement of ulceration at the nasal mucosa at the discretion of the investigator (yes or no)
Pain at sensor insertion site | 7 days
  Pain at the insertion site measured by Numeric Rating Scale (0= no pain, 10= maximum pain)

OTHER OUTCOMES:
Muscular temperature level | 14 hours
  Muscular temperature level (grade Celsius) during insertion period
Nasal temperature level | 14 hours
  Nasal temperature level (grade Celsius) during insertion period
Temporal temperature level | 14 hours
  Temporal temperature level (grade Celsius) during insertion period
IscAlert functionality | 14 hours
  Number of hours with a well-functioning sensor (giving carbon dioxide- and temperature data)
Number of pack-years | 7 days
  Smoking habit; number of pack-years by participants
Length of sensor implantation time | 7 days
  Length of sensor implantation time during hospitalisation
Peripheral oxygen saturation | 14 hours
  Peripheral oxygen saturation (SpO2)
Arterial partial pressure (level) of carbon dioxide | 14 hours
  Arterial partial pressure of carbon dioxide (kPa) during insertion period - measured in arterial blood
Arterial partial pressure (level) of oxygen | 14 hours
  Arterial partial pressure of oxygen (kPa) during insertion period - measured in arterial blood
Intramuscular partial pressure (level) of carbon dioxide | 14 hours
  Intramuscular partial pressure of carbon dioxide (kPa) during insertion period - measured in the forearm
Transcutaneous partial pressure (level) of carbon dioxide | 14 hours
  Transcutaneous partial pressure of carbon dioxide (kPa) during insertion period, measured at the skin of the forehead
Patient-Reported Outcome Measures 1a - discomfort | 14 hours
  Discomfort in the nose - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 1b - discomfort | 7 days
  Discomfort in the nose - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 2a - runny nose | 14 hours
  Runny nose - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 2b - runny nose | 7 days
  Runny nose - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 3a - sneezing | 14 hours
  Sneezing - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 3b - sneezing | 7 days
  Sneezing - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 3b - Ulceration | 7 days
  Ulceration in the nose mucouse membrane - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 3a - Ulceration | 14 hours
  Ulceration in the nose mucouse membrane - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 4a - tenderness | 14 hours
  Tenderness in the nose - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 4b - tenderness | 7 days
  Tenderness in the nose - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 5b - bleeding | 7 days
  Bleeding from the nose - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 5a - bleeding | 14 hours
  Bleeding from the nose - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 6a - reduced sense of smell | 14 hours
  Reduced sense of smell - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 6b - reduced sense of smell | 7 days
  Reduced sense of smell - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 7b - reduced sense of taste | 7 days
  reduced sense of taste - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 7a - reduced sense of taste | 14 hours
  reduced sense of taste - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 8a - difficulty sleeping | 14 hours
  difficulty sleeping - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 8b - easy to wake up while sleeping | 7 days
  easy to wake up while sleeping - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 9 - problems with eating and drinking | 14 hours
  problems with eating and drinking - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 10 - difficult breathing | 14 hours
  difficult breathing - Patient-Reported Outcome Measure, Scale 1 to 5 (1= no, 2= little, 3=Some, 4=very 5=Extreme)
Patient-Reported Outcome Measures 11a - diagnosed infection in the nose or sinuses | 14 hours
  diagnosed infection in the nose or sinuses - Patient-Reported Outcome Measure, Scale 1 to 2 (1= No, 2= Yes)
Patient-Reported Outcome Measures 11b - diagnosed infection in the nose or sinuses | 7 days
  diagnosed infection in the nose or sinuses - Patient-Reported Outcome Measure, Scale 1 to 2 (1= No, 2= Yes)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Gabrielsen, MD, PhD, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Vestfold Hopsital Trust, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD to other researchers